CLINICAL TRIAL: NCT00002887
Title: PHASE I TRIAL OF HYDROXYUREA FOR SALVAGE OF INCURABLE NON-SMALL CELL LUNG CANCER
Brief Title: Hydroxyurea Plus Combination Chemotherapy in Patients With Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Regional Cancer Centre (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065207; CAN-OTT-9501; NCI-V96-1099
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-10

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Etoposide; Hydroxyurea; Vinblastine; Vindesine; Vinorelbine

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Drug: hydroxyurea
Drug: vinblastine sulfate
Drug: vindesine
Drug: vinorelbine tartrate
Procedure: drug resistance inhibition treatment

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug is a way to kill more tumor cells.

PURPOSE: Phase I trial to study the effects of hydroxyurea plus combination chemotherapy in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the maximum tolerated dose of hydroxyurea that can be given in combination with other chemotherapy regimens in patients with incurable non-small cell lung cancer. II. Determine the toxicity of this combination chemotherapy regimen in these patients. III. Observe the efficacy of hydroxyurea in patients with incurable non-small cell lung cancer refractory to front-line chemotherapy.

OUTLINE: This study seeks to estimate the maximum tolerated dose (MTD) of hydroxyurea in combination with other chemotherapy. Groups of 3 patients take escalated doses of oral hydroxyurea three times weekly or daily throughout treatment with cisplatin plus (per their previous regimen) vinblastine, vindesine, vinorelbine, or etoposide. Treatment continues in responding and stable patients until 3 months beyond documentation of complete remission (minimum 4 courses), maximum of 6 courses beyond documentation of partial remission, or 3 courses beyond documentation of stable disease. Patients are followed every 3 weeks for 3 months, every 6 weeks for 3 months, then every 3 months until disease progression.

PROJECTED ACCRUAL: An anticipated 15-30 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histopathologically proven non-small cell lung cancer that is incurable by surgery or radiotherapy Brain metastases allowed Demonstrated resistance to prior chemotherapy required by 1 of the following: Tumor growth or recurrence while on treatment Failure of tumor to shrink over 3 consecutive courses of treatment Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: ANC at least 1,500 Platelets at least 100,000 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 1.5 mg/dL (26 micromoles/L) AST/ALT less than 1.5 times normal Renal: Creatinine less than 1.6 mg/dL (150 micromoles/L) Cardiovascular: No uncontrolled hypertension or other cardiac disease No myocardial infarction within 6 months Other: No uncontrolled diabetes No active abuse of ethanol No allergies to study medication No active infection or other serious medical condition that precludes protocol treatment No dementia or significantly altered mental status that precludes informed consent No prior melanoma or malignancy of the following sites: Breast Kidney Thyroid Salivary glands Endometrium No other second malignancy within 5 years except: Nonmelanomatous skin cancer Carcinoma in situ of cervix No pregnant or nursing women Effective contraception required of fertile women

PRIOR CONCURRENT THERAPY: Recovery from any treatment-limiting toxicity required Biologic therapy: Not specified Chemotherapy: At least 3 weeks since myelosuppressive chemotherapy (6 weeks since nitrosoureas, mitomycin, or high-dose carboplatin) Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since radiotherapy unless to a limb or limited treatment area Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Overall Officials: David J. Stewart, MD, FRCPC, Study Chair — Ottawa Regional Cancer Centre
Locations (1):
- Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario, Canada